CLINICAL TRIAL: NCT03937609
Title: Randomized, Multicenter Study to Investigate the Efficacy of Dashboard Driven Individualized Dosing of Infliximab Compared To Standard Dosing During the Induction in Patients With Acute Severe Ulcerative Colitis
Brief Title: TITRATE (inducTIon for acuTe ulceRATivE Colitis)
Acronym: TITRATE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Geert D'Haens, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6746101818
Record Dates: First submitted 2019-04-30; First posted 2019-05-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Colitis, Ulcerative
Keywords: infliximab
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Infliximab; CT-P13

STUDY DESIGN:
Intervention Model Description: Randomized, Open-label, Multicenter Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard dosing (Other): All eligible patients will receive an intravenous infusion of IFX at 5 mg/kg IFX at week 0. The control group will continue with 5 mg/kg IFX at week 2 and 6, followed by every 8 weeks.
  Interventions: Drug: Infliximab
- Intervention group (Experimental): All eligible patients will receive an intravenous infusion of IFX at 5 mg/kg IFX at week 0. The intervention group will receive model based dosing of infliximab with 5mg/kg at various timepoints based on the dashboard model.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — infliximab iv 5mg/kg
  Other Names: Remicade, Inflectra and Remsima

SUMMARY:
The aim of this study is to investigate whether intensive, personalized IFX dosing by using a pharmacokinetics driven dashboard system during the induction phase in patients with acute severe UC leads to increased treatment success (as defined by clinical and endoscopic response at week 6) as compared to the standard dosing.

DETAILED DESCRIPTION:
Previous studies performed in the AMC demonstrated that the patients with acute severe UC receiving IFX are different from patients receiving IFX while in remission.(5) The clearance of IFX is not only determined by demographic parameters (gender, body weight), blood chemistry (CRP, albumin) and anti-drug antibodies, but also disease related variables play an important role. Among others, we have demonstrated that faecal loss of IFX in ASUC patients increases IFX clearance during the induction phase (3). Furthermore, increased expression of TNF-α, the target of IFX, influences the clearance of IFX due to target mediated drug disposition (TMDD). Active IBD with high tissue concentrations of TNF-α thereby acts as a sink for anti-TNF-α antibodies (4). The PK of IFX has been mainly characterized during maintenance therapy. Evaluation of factors that influence the clearance of IFX during induction therapy will allow further optimization an individualization of IFX therapy in ASUC patients.

At present, determination of IFX concentrations in the serum with an enzyme-linked immunosorbent assay (ELISA) is time consuming; physicians often receive the results after as many as 10-20 days. To allow for proactive adjustments in dosing, faster laboratory results are required, preferably in a point-of-care setting. This test is now made available by Bühlmann Laboratories (Switzerland).

The study hypothesis is that in patients with acute severe UC an intensified and personalized IFX dosing regimen using individual PK data from point of care tests as a rapid input to the dashboard system during the induction phase will lead to improved clinical outcomes when compared to standard dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Admission with acute severe UC (defined patients with bloody diarrhoea ≥ 6/day and any signs of systemic toxicity (pulse > 90/min, temperature > 37.8°C, haemoglobin < 105 g/l, erythrocyte sedimentation rate [ESR] > 30 mm/h, or C-reactive protein [CRP] > 30 mg/l)
2. Failure to intravenous steroid treatment as defined by the Oxford criteria (more than 8 stools/d or 3-8 stools/d and CRP≥45) and a Lichtiger score ≥ 10 on day 3 after starting iv steroid treatment
3. Patients going through baseline endoscopy and biopsy sampling (including CMV) before starting on IFX treatment
4. In the opinion of the investigator, the subject is capable of understanding and complying with protocol requirements.
5. The subject signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
6. Male or non-pregnant, non-lactating females. Females of child bearing potential must have a negative serum pregnancy test prior to randomization, and must use a hormonal (oral, implantable or injectable) or barrier method of birth control throughout week 26. Females unable to bear children must have documentation of such in the source records (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]).

Exclusion Criteria:

1. Patients at imminent need of surgery as judged by the treating clinician
2. Previous use of IFX
3. Enteric pathogens (such as Salmonella, Shigella, Yershinia, Campylobacter and C. difficile) detected by stool analysis within 2 weeks prior to enrollment or at screening
4. Active participation in another interventional trial
5. Patients with Crohn's disease or IBD-U
6. Patients with abdominal abscess
7. Patients with colonic stricture
8. Patients with a history of colon cancer or colonic dysplasia, unless sporadic adenoma, which has been removed
9. Active or latent tuberculosis (screening according to national guidelines)
10. Cardiac failure in NYHA stage III-IV
11. History of demyelinating disease
12. Recent live vaccination
13. Patients with ongoing acute/chronic infection (including but not limited to HIV, hepatitis B and C) with the exception of chronic herpes labialis or cervical HPV
14. History of cancer in the last 5 years with the exception of non-melanoma skin cancer
15. A history of alcohol or illicit drug use that in the opinion of the principal investigator (PI) would interfere with study procedures
16. Patients with psychiatric problems that in the opinion of the PI would interfere with study procedures
17. Patients unable to attend all study visits
18. Patients with a history of non-compliance with clinical study protocols
19. Contraindication for endoscopy
20. Patients who received any investigational drug in the past 30 days or 5 half-lives, whichever is longer
21. Patients who received cyclosporine in the previous 14 days
22. Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Increased treatment success | week 6
  Defined by clinical and endoscopic reponse. Clinical response defined as a Lichtiger score of less than 10 points with a decrease of at least 3 points compared to baseline. Endoscopic response is defined as a decrease of at least 2 points in the UCEIS at week 6 endoscopy compared to baseline

SECONDARY OUTCOMES:
Endoscopic Remission | week 6 and week 26
  Mayo score 2 or less with no individual subscore less than 1
Endoscopic Reponse | week 6 and week 26
  Decrease in Mayo score of 3 or more points and a 30% or more from baseline and a decrease in rectal bleeding score of 1 or more or an absolute rectal bleeding score of 0 or 1
Clinical Remission | Week 6 and week 26
  Measured by the Simple Clinical Colitis Activity Index (SCCAI score ≤ 2)
Corticosteroid-free remission | week 26
  Measured by the Simple Clinical Colitis Activity Index (SCCAI score ≤ 2)

CONTACTS AND LOCATIONS:
Overall Officials: Geert DHaens, Principal Investigator — Amsterdamumc location AMC
Locations (7):
- St Vincent's University Hospital, Dublin, Ireland
- Netherlands (3):
  - Academic Medical Center, Amsterdam
  - OLVG Oost, Amsterdam
  - Radboud UMC, Nijmegen
- Norway (3):
  - Klinikk Baerum Sykehus, Bærums verk
  - Akerhus University Hospital, Lørenskog
  - Helse Stavanger, Stavanger

IPD SHARING:
Plan to Share IPD: No